CLINICAL TRIAL: NCT00968435
Title: Phase II Trial of Bevacizumab, Cetuximab, and Cisplatin With IMRT (Intensity-Modulated Radiation Therapy) for Patients With Stage III/IV Head and Neck Squamous Cell Carcinoma
Brief Title: Bevacizumab, Cetuximab, and Cisplatin With IMRT (Intensity-Modulated Radiation Therapy) for Patients With Stage III/IV Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-083
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Head and Neck Cancer
Keywords: bevacizumab; cisplatin; cetuximab; radiation therapy; Phase II; 09-083
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Bevacizumab; Cisplatin; Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (IMRT) + cisplatin + bevacizumab + cetuximab (Experimental): This is a single-institution, non-randomized, phase II study. The primary endpoint is to determine 2-year progression-free survival for patients with locally or regionally advanced HNSCC treated with concurrent intensity modulated radiation therapy (IMRT) + cisplatin + bevacizumab + cetuximab.
  Interventions: Other: bevacizumab, cisplatin, cetuximab, radiation therapy

INTERVENTIONS:
Other: bevacizumab, cisplatin, cetuximab, radiation therapy — Patients will receive intensity-modulated radiation therapy (IMRT) in once-daily fractions. A total dose of 70Gy is planned for the primary tumor site over approximately 33 treatment days. Day 1 will refer to the first day of radiation therapy. Concurrent with radiation therapy, patients will receive cisplatin (50 mg/m2 IV on Days 1, 2 and 22, 23) and bevacizumab (15 mg/kg IV on Days 1 and 22). Cetuximab will be administered according to the Bonner regimen (4),with a loading dose approximately 7 days prior to the start of radiation therapy (400 mg/m2 IV once, on approximately Day minus 7), followed by weekly cetuximab infusions (250 mg/m2 IV weekly X 7 infusions) until the completion of radiation therapy.

SUMMARY:
The purpose of this study is to determine the effectiveness of treatment with bevacizumab + cisplatin + cetuximab + IMRT. The doctor wishes to monitor patients for 2 years after the completion of study treatment to determine if they are cancer-free during that time. They also want to evaluate the side effects that patients experience with this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Stage III/IV HNSCC without distant metastasis. Patients with stage II squamous cell carcinoma of the hypopharynx will also be eligible
* Adequate renal function, with serum creatinine ≤ 1.5 mg/dL. Patients with serum creatinine > 1.5 mg/dL may be eligible if calculated creatinine clearance > or = to 55 ml/min by Cockcroft and Gault equation (or 24-hour urine collection).
* Age > or = to 18 years.
* Karnofsky performance status > or = to 70%
* Adequate bone marrow function: absolute neutrophil count > or = to 1,500/ platelets > or = to 100,000/ul, hemoglobin > or = to 9 gm/dl
* Adequate hepatic function: Total bilirubin ≤ 1.5 X ULN (patients with Gilbert's syndrome as the cause of hyperbilirubinemia may be eligible if total bilirubin ≤ 2.5 X ULN), aspartate aminotransferase (AST) ≤ 2.5 X ULN, alanine aminotransferase (ALT) ≤ 2.5 X ULN, alkaline phosphatase ≤ 2.5 X ULN.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation therapy for HNSCC
* Prior treatment of HNSCC with bevacizumab or other agents specifically targeting VEGF
* Prior treatment of HNSCC with cetuximab or other agents specifically targeting EGFR
* Other active malignancy, other than indolent malignancies, which the investigator determines are unlikely to interfere with treatment or efficacy analysis. For example, patients with non-melanoma skin cancer, in situ carcinoma of the cervix, or prostate cancer within the no current biochemical (PSA) or radiologic evidence of disease may enroll.
* Patients with nasopharyngeal carcinoma
* Patients who will receive amifostine as part of the radiation treatment plan
* Patients with skin breakdown/ulceration (CTCAE version 3.0, grade 2 or higher).
* Patients with hearing loss requiring hearing aid or intervention (i.e. interfering in a clinically significant way with activities of daily living).
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living).
* Any prior documented history of transient ischemic attack (TIA) or cerebrovascular accident (CVA)
* History of unstable angina or myocardial infarction (MI) within the last year.
* Urine protein: creatinine (UPC) ratio > or = to 1.0 at screening. A random urine sample is collected. Total protein (mg/dL) and spot creatinine (mg/dL) are ordered for this sample. The UPC ratio is calculated from the results of these tests.
* International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (aPTT) > 1.5 X upper limits of normal (ULN)
* Current use of warfarin, current use of heparin or low-molecular weight heparin, chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function.
* Patients with gross hemoptysis or hematemesis (defined as bright red blood of 1 teaspoon of more) within 28 days prior to Day 0 protocol treatment will be excluded from this trial. Patients with incidental blood mixed with phlegm are not excluded.
* Esophageal varices, non-healing ulcer, wound, or bone fracture are exclusion criteria. However, patients with skin breakdown overlying malignant neck lymphadenopathy may be eligible, at the discretion of the investigator.
* Anatomic lesion that increases the risk of serious hemorrhage, such as encasement or invasion of major blood vessels by primary tumor and/or by involved lymph nodes
* Blood pressure of > 150/100 mmHg
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* Clinically significant peripheral vascular disease
* History of bleeding diathesis or hemorrhagic disorder, or coagulopathy.
* Major surgical procedure or significant traumatic injury within 28 days prior to treatment with bevacizumab
* Core biopsy within 7 days prior to treatment with bevacizumab.
* Minor surgical procedures such as fine needle aspirations or placement of percutaneous gastrostomy tube (PEG) less than 7 days prior to treatment with bevacizumab
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior enrollment.
* Inability to comply with study and/or follow-up procedures
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To determine the 2-year progression-free survival for patients with locally or regionally advanced HNSCC treated with concurrent IMRT + cisplatin + bevacizumab + cetuximab. | 2 years

SECONDARY OUTCOMES:
To determine median overall survival for patients with locally or regionally advanced HNSCC treated with concurrent IMRT + cisplatin + bevacizumab + cetuximab. | 2 years
To evaluate the safety and tolerability of concurrent IMRT + cisplatin + bevacizumab + cetuximab. | 2 years
To explore the potential utility of 18F FLT PET for early response assessment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm